CLINICAL TRIAL: NCT05779046
Title: The Acute Effect of High Intensity Interval Exercise on Respiratory Function and Rhinitis Symptoms in Patients With Allergic Rhinitis
Brief Title: Acute Effect of High Intensity Interval Exercise in Patients With Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wannaporn Tongtako, Ph.D., Principal investigator, Chulalongkorn University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EX PHYSIO SPSC 5
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinits; Acute exercise; High intensity interval training; Rhinitis symptoms; nasal blood flow
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Twelve patients with allergic rhinitis aged between 19 and 31 years who had a positive skin prick test to house dust mite (D. pteronyssinus). The experiment was a crossover design in which each participant was given two types of high-intensity interval training exercise (HIT): HIT 1:1 (high intensity for 1 minute at 85-90% of maximum heart rate, then alternating with low intensity 50-55% of maximum heart rate for 1 minute) and HIT 1:2 (high intensity for 1 minute at 85-90% of maximum heart rate, then alternating with low intensity 50-55% of maximum heart rate for 2 minutes). Rhinitis symptoms, nasal blood flow, peak nasal inspiratory flow, pulmonary functions, respiratory muscle strength, and fractional exhaled nitric oxide were measured before and immediately, 15 minutes, 30 minutes, 45 minutes, and 60 minutes after exercise for each exercise program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIT 1:1 (Experimental): The participants received a high-intensity interval exercise program of walking or running on a treadmill for approximately 40 minutes. The training included a 10-minute warm-up at low intensity. High-intensity interval exercise at a ratio of 1:1 (high intensity for 1 minute at 85-90% of maximum heart rate, then alternating with low intensity 50-55% of maximum heart rate for 1 minute ).
  Interventions: Other: HIT 1:1
- HIT 1:2 (Experimental): The participants received a high-intensity interval exercise program of walking or running on a treadmill for approximately 40 minutes. The training included a 10-minute warm-up at low intensity. High-intensity interval exercise at a ratio of 1:2 (high intensity for 1 minute at 85-90% of maximum heart rate, then alternate with low intensity 50-55% of maximum heart rate for 2 minutes).
  Interventions: Other: HIT 1:2

INTERVENTIONS:
Other: HIT 1:1 — The participants received a high-intensity interval exercise program of walking or running on a treadmill for approximately 40 minutes. The training included a 10-minute warm-up at low intensity. High-intensity interval exercise at a ratio of 1:1 (high intensity for 1 minute at 85-90% of maximum heart rate, then alternating with low intensity 50-55% of maximum heart rate for 1 minute).
  Arms: HIT 1:1
Other: HIT 1:2 — The participants received a high-intensity interval exercise program of walking or running on a treadmill for approximately 40 minutes. The training included a 10-minute warm-up at low intensity. High-intensity interval exercise at a ratio of 1:2 (high intensity for 1 minute at 85-90% of maximum heart rate, then alternate with low intensity 50-55% of maximum heart rate for 2 minutes).
  Arms: HIT 1:2

SUMMARY:
The purpose of this study was to determine the acute effect of high intensity interval exercise on respiratory function and rhinitis symptoms in allergic rhinitis patients.

DETAILED DESCRIPTION:
Twelve patients with allergic rhinitis aged between 19 and 31 years who had a positive skin prick test to house dust mite (D. pteronyssinus). The experiment was a crossover design in which each participant was given two types of high-intensity interval training exercise (HIT): HIT 1:1 (high intensity for 1 minute at 85-90% of maximum heart rate, then alternating with low intensity 50-55% of maximum heart rate for 1 minute) and HIT 1:2 (high intensity for 1 minute at 85-90% of maximum heart rate, then alternating with low intensity 50-55% of maximum heart rate for 2 minutes). Rhinitis symptoms, nasal blood flow, peak nasal inspiratory flow, pulmonary functions, respiratory muscle strength, and fractional exhaled nitric oxide were measured before and immediately, 15 minutes, 30 minutes, 45 minutes, and 60 minutes after exercise for each exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Subjects had a clinical history of persistent rhinitis, and had positive skin prick test to house dust mite (D. pteronyssinus)
* Persistent allergic rhinitis
* Subjects with known asthma, chronic rhinosinusitis, Lung cancer and Emphysema diseases were excluded.
* BMI 18.5 - 24.9 kg/m2
* Subjects will ask to abstain from taking antihistamine for at least 5 days, leukotriene receptor antagonist for at least 1 week, and nasal steroids for at least 2 weeks prior to the start of the experiment.
* Subjects will ask to abstain from taking any form of dietary supplement during the experiment.
* Subjects had no exercise training program (not exercise regularly or not exercise for 30 minutes or more at least 3 times per week during the past 6 months)

Exclusion Criteria:

* Accident that are unable to continue the research, such as accidental injury or illness, etc.
* Participants did not voluntarily participate.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Rhinitis symptom scores change | Change after each exercise immediately, 15 minutes, 30 minutes, 45 minutes, and 60 minutes
  Nasal symptoms were assessed using Total Nasal Symptom Score (TNSS) questionnaire. The subjects were asked to score symptoms of persistent allergic rhinitis before and after yoga training protocol. The total nasal symptom scores were computed as the sum of four individual nasal symptom scores; nasal congestion, itching, sneezing, and rhinorrhea. The scores ranged from 0 to 3 scale (0=none, 1=mild, 2=moderate, 3= severe)
Peak nasal inspiratory flow change | Change after each exercise immediately, 15 minutes, 30 minutes, 45 minutes, and 60 minutes
  The subjects placed a mask, which is turned onto a plastic cylinder through which the air passes during inspiration, over the nose and mouth and inspired forcefully through the nose, with lips tightly closed. Inside the cylinder, there is a diaphragm that moves to the airflow, and the maximum peak flow is registered in a scale range from 30-370 L/min. During the procedure, the subjects placed a mask over the nose and mouth and inspired forcefully through the nose, with lips tightly closed.
Nasal blood flow change | Change after each exercise immediately, 15 minutes, 30 minutes, 45 minutes, and 60 minutes
  Laser Doppler flowmetry (DRT4 moor instrument, UK.) was used to measure of the nasal blood flow (NBF). Before the test each subject rested for one hour in a separate room. During the test, they were instructed to breathe normally breathe and not to speak, cough, or move. A lateral endoscopic probe with a flexible nylon sheath 1.34-mm-diameter flexible nylon sheath was placed to the front of the nose. Nasal blood flow measurements were performed before immediately, 15 minutes, 30 minutes, 45 minutes, and 60 minutes after exercise for each exercise program.
Pulmonary functions change | Change after each exercise immediately, 15 minutes, 30 minutes, 45 minutes, and 60 minutes
  The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration.
Respiratory muscle strength change | Change after each exercise immediately, 15 minutes, 30 minutes, 45 minutes, and 60 minutes
  Respiratory muscle strength was assessed by measuring Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) in cmH2O. The participants were in a sitting position using a portable handheld mouth pressure meter (i.e., MicroRPM) with a nose clip. For the MIP measurement, the participants were asked to exhale until they felt no air remaining in their lungs (starting with the functional residual capacity [FRC] point), then held the device on their mouth and inhaled forcefully for 1-2 seconds. For the MEP measurement, the participants were asked to inhale until their lungs were completely filled with air (starting with the total lung capacity [TLC] point), then they kept the device on their mouth and exhaled forcefully for 1-2 seconds

SECONDARY OUTCOMES:
Fractional exhaled nitric oxide | Change after each exercise immediately, 15 minutes, 30 minutes, 45 minutes, and 60 minutes
  Participants inhaled deeply for two to three seconds before exhaling slowly. Normally, it took 10 seconds to exhale.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

REFERENCES:
- [Background] Savoure M, Bousquet J, Jaakkola JJK, Jaakkola MS, Jacquemin B, Nadif R. Worldwide prevalence of rhinitis in adults: A review of definitions and temporal evolution. Clin Transl Allergy. 2022 Mar;12(3):e12130. doi: 10.1002/clt2.12130. PMID 35344304
- [Background] Min YG. The pathophysiology, diagnosis and treatment of allergic rhinitis. Allergy Asthma Immunol Res. 2010 Apr;2(2):65-76. doi: 10.4168/aair.2010.2.2.65. Epub 2010 Mar 24. PMID 20358020
- [Background] Kalpaklioglu AF, Kalkan IK. Comparison of orally exhaled nitric oxide in allergic versus nonallergic rhinitis. Am J Rhinol Allergy. 2012 Mar-Apr;26(2):e50-4. doi: 10.2500/ajra.2012.26.3717. PMID 22487277
- [Background] Tongtako W, Klaewsongkram J, Jaronsukwimal N, Buranapraditkun S, Mickleborough TD, Suksom D. The effect of acute exhaustive and moderate intensity exercises on nasal cytokine secretion and clinical symptoms in allergic rhinitis patients. Asian Pac J Allergy Immunol. 2012 Sep;30(3):185-92. PMID 23156847
- [Background] Dunham C, Harms CA. Effects of high-intensity interval training on pulmonary function. Eur J Appl Physiol. 2012 Aug;112(8):3061-8. doi: 10.1007/s00421-011-2285-5. Epub 2011 Dec 23. PMID 22194005
- [Background] Andrade DC, Arce-Alvarez A, Parada F, Uribe S, Gordillo P, Dupre A, Ojeda C, Palumbo F, Castro G, Vasquez-Munoz M, Del Rio R, Ramirez-Campillo R, Izquierdo M. Acute effects of high-intensity interval training session and endurance exercise on pulmonary function and cardiorespiratory coupling. Physiol Rep. 2020 Aug;8(15):e14455. doi: 10.14814/phy2.14455. PMID 32748551
- [Background] Gao M, Huang Y, Wang Q, Liu K, Sun G. Effects of High-Intensity Interval Training on Pulmonary Function and Exercise Capacity in Individuals with Chronic Obstructive Pulmonary Disease: A Meta-Analysis and Systematic Review. Adv Ther. 2022 Jan;39(1):94-116. doi: 10.1007/s12325-021-01920-6. Epub 2021 Nov 18. PMID 34792785